CLINICAL TRIAL: NCT04364542
Title: Suprascapular Nerve Block Efficacy for Arthroscopic Rotator Cuff Repair: a Randomized Clinical Trial
Brief Title: Suprascapular Nerve Block Efficacy for Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ivan Simionato (Other)
Responsible Party: Sponsor-Investigator, Ivan Simionato, Clinical Researcher, Shoulder Surgery Group, Santa Casa de Porto Alegre
Organization: Shoulder Surgery Group, Santa Casa de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShoulderSurgeryGroupSCPA
Record Dates: First submitted 2020-03-11; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Shoulder Pain; Postoperative Pain; Rotator Cuff Tears; Anesthesia; Anesthesia, Local
Keywords: Shoulder surgery; Pain; Brachial plexus blockage; Anesthesia; Interscalene blockage; Opioid
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Rotator Cuff Injuries; Pain

STUDY DESIGN:
Intervention Model Description: 2 groups of patients. Randomization into groups SSNB or ISB as per randomization list, for a total of 98 patients
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, and Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprascapular nerve block (SSNB) (Experimental): Single shot using the blind block technique with 10 ml 0.75% ropivacaine and arthroscopic portals infiltration with 5 ml 0.75% diluted in 15 ml of distilled water.
  Interventions: Procedure: Suprascapular nerve block; Procedure: Arthroscopic rotator cuff repair
- Interscalene Nerve Block (ISB) (Active Comparator): Single shot using US-guided interscalene brachial plexus block with 15 ml 0.5% ropivacaine and arthroscopic portals infiltration with 5 ml 0.75% diluted in 15 ml of distilled water.
  Interventions: Procedure: Interscalene Nerve Block; Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Suprascapular nerve block — The patient lies supine in beach chair position with surgical drapes on. The anatomical landmarks are outlined and the infiltration spot is identified. The block is performed with 10 ml ropivacaine 0.75%.
  Arms: Suprascapular nerve block (SSNB)
Procedure: Interscalene Nerve Block — The patient lies supine position with the head turned to the contralateral side to the block. A linear high-frequency ultrasound probe is used for identifying the roots of supraclavicular brachial plexus using the traceback technique. The block is performed with 15 ml ropivacaine 0.5%.
  Other Names: Interscalene Brachial Plexus Nerve Blockade
  Arms: Interscalene Nerve Block (ISB)
Procedure: Arthroscopic rotator cuff repair — Conventional arthroscopic rotator cuff repair.

SUMMARY:
This study evaluates the analgesia induced by suprascapular nerve block in comparison to interscalene nerve block in arthroscopic rotator cuff repairs. The experimental and the control group will receive the suprascapular nerve block and interscalene nerve block, respectively.

DETAILED DESCRIPTION:
Peripheral nerve blocks are widely used for postsurgical analgesia. Interscalene nerve block provides a total brachial plexus motor and sensitive blockade while the suprascapular nerve block produces only a specific peripheral blockade.

The interscalene nerve block is the most frequently used anesthesia technique and requires a longer learning curve. Complications related to this technique may be more severe and frequent in comparison to other regional anesthesia techniques.

The suprascapular nerve block yields less adverse effects, discomfort and rebound effect as this technique does not completely block the upper limb motor function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Confirmed rotator cuff tear by magnetic resonance imaging

Exclusion Criteria:

* Irreparable cuff tears (retracted lesions to the glenoid rim and/or fourth grade fatty infiltration)
* Partial repair of cuff tears (immobile lesions)
* Rheumatic diseases
* Neck-related shoulder pain
* Glenohumeral instability or osteoarthritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: Numeric Pain Rating Scale | 1 hour after surgery
  Numeric Pain Rating Scale - no pain (0), unbearable pain (10)
Pain intensity: Numeric Pain Rating Scale | 24 hours after surgery
  Numeric Pain Rating Scale - no pain (0), unbearable pain (10)
Pain intensity: Numeric Pain Rating Scale | 48 hours after surgery
  Numeric Pain Rating Scale - no pain (0), unbearable pain (10)
Pain intensity: Numeric Pain Rating Scale | 72 hours after surgery
  Numeric Pain Rating Scale - no pain (0), unbearable pain (10)

SECONDARY OUTCOMES:
Opiate Consumption | Postoperative hours 1-72
  Total amount of narcotics consumed during the postoperative period measured in morphine equivalents (OME).

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Silva, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Background] Lindberg MF, Grov EK, Gay CL, Rustoen T, Granheim TI, Amlie E, Lerdal A. Pain characteristics and self-rated health after elective orthopaedic surgery - a cross-sectional survey. J Clin Nurs. 2013 May;22(9-10):1242-53. doi: 10.1111/jocn.12149. Epub 2013 Mar 29. PMID 23551432
- [Background] Desai N. Postoperative analgesia for shoulder surgery. Br J Hosp Med (Lond). 2017 Sep 2;78(9):511-515. doi: 10.12968/hmed.2017.78.9.511. PMID 28898151
- [Background] Hussain N, Goldar G, Ragina N, Banfield L, Laffey JG, Abdallah FW. Suprascapular and Interscalene Nerve Block for Shoulder Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2017 Dec;127(6):998-1013. doi: 10.1097/ALN.0000000000001894. PMID 28968280
- [Background] Vandepitte C, Gautier P, Xu D, Salviz EA, Hadzic A. Effective volume of ropivacaine 0.75% through a catheter required for interscalene brachial plexus blockade. Anesthesiology. 2013 Apr;118(4):863-7. doi: 10.1097/ALN.0b013e3182850dc7. PMID 23353796
- [Background] Lee JJ, Kim DY, Hwang JT, Lee SS, Hwang SM, Kim GH, Jo YG. Effect of ultrasonographically guided axillary nerve block combined with suprascapular nerve block in arthroscopic rotator cuff repair: a randomized controlled trial. Arthroscopy. 2014 Aug;30(8):906-14. doi: 10.1016/j.arthro.2014.03.014. Epub 2014 May 29. PMID 24880194
- [Background] Toma O, Persoons B, Pogatzki-Zahn E, Van de Velde M, Joshi GP; PROSPECT Working Group collaborators. PROSPECT guideline for rotator cuff repair surgery: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2019 Oct;74(10):1320-1331. doi: 10.1111/anae.14796. Epub 2019 Aug 7. PMID 31392721